CLINICAL TRIAL: NCT07018219
Title: Identification of the Seventh Cervical Vertebra by Palpation With Neck Rotation and Side Bending in Patients With Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eslam Elsayed Ali Shohda (Other Government)
Responsible Party: Sponsor-Investigator, Eslam Elsayed Ali Shohda, Physical therapy teaching fellow, General Committee of Teaching Hospitals and Institutes, Egypt
Organization: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HAH00059
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: Identification of the Seventh Cervical Vertebra by Palpation
Keywords: Seventh Cervical vertebra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one expermental group: (Experimental): The researcher will detect the seventh cervical vertebrae by palpation with neck Rotation and side bending in patients with neck pain , then patients will be refereed to perform X ray which is the gold standard for detecting C7
  Interventions: Device: X ray device

INTERVENTIONS:
Device: X ray device — X ray macjine : shimadzo corporation ( japan)

SUMMARY:
detect accuracy of that procedure in identification the seventh cervical vertebra, we aimed to determine accuracy of identification of the seventh cervical vertebra by palpation with neck rotation and side bending in patients with neck pain.

DETAILED DESCRIPTION:
The ability to identify the correct vertebral level through examination is an important skill for clinicians in many different specialities (1,2). Two methods for identifying seventh cervical vertebra are commonly used; the conventional palpation method, which identifies the most prominent cervical spinous process as the seventh cervical (C7) spinous process and flexion-extension method which identifies the lowest freely moving spinous process as C6 and the following stationary cervical spinous process as C7. One study found the accuracy of the conventional palpation method is 37.5% while the accuracy of the flexion-extension is 77.1%. Another method is done by detecting the most prominent three vertebrae at cervicothoracic junction then three palpating fingers will be placed paravertebrally to the left of the cervicothoracic region against the left side of the assumed C7 and Tl spinous processes. When rotation or lateral flexion is facilitated, C7 is expected to move significantly further than the more slowly reacting Tl spinous process.

ELIGIBILITY:
Inclusion Criteria:

* neck pain, age (18- 60) male and female

Exclusion Criteria:

* with suspected ankylosing spondylitis, previous surgery on the cervical spine or congenital malformation of the cervical region.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-03 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
The accuracy of palpation technique | 2 month
  The accuracy of palpation technique will be calculated as the proportion of patients in which the palpated vertebral level corresponded to the radiographic vertebral level.

CONTACTS AND LOCATIONS:
Locations (1):
- Al ahrar teaching hospital, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
undetected